CLINICAL TRIAL: NCT01188720
Title: Sexual Health on Antidepressants Through Physical Exercise
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tierney Kyle Ahrold Lorenz, Researcher, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-07-0043; F31MH085416 (NIH)
Record Dates: First submitted 2010-08-20; First posted 2010-08-25 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baseline (No Intervention): Assessment only baseline
- Acute exercise (Experimental): Exercise immediately before sexual activity, three times per week.
  Interventions: Behavioral: Physical activity
- General exercise (Active Comparator): Exercise not immediately before sexual activity, three times per week.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — 30 minutes of moderate to intense physical activity including strength training and cardiovascular activity.
  Arms: Acute exercise; General exercise

SUMMARY:
Preliminary findings from a trial in the investigators laboratory suggest that acute exercise may ameliorate deficits in sexual arousal associated with use of antidepressants. The goal of this project is to evaluate the real-world effectiveness of an exercise-based intervention for these side effects in a community-based sample. The investigators hypothesize that general exercise will help improve sexual functioning in women taking antidepressants, and that exercise immediately before sexual activity - that is, acute exercise - will have an additional beneficial effect above and beyond that of general exercise.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 18 or older
* currently receiving a consistent dosage of escitalopram, citalopram, sertraline, desvenlafaxine, venlafaxine, or duloxetine
* currently sexually active
* willing and able to exercise
* experiencing regular menstrual cycles
* not currently pregnant and not intending to become pregnant during trial

Exclusion Criteria:

* currently taking more than one psychoactive medication
* factors indicating risk of cardiovascular activity, including acute or chronic cardiovascular illness, including clinically significant hypertension (defined as self-reported hypertension or "blood pressure greater than 140/90" or receiving medications designed to treat hypertension); recent chest pain; frequent or recurrent faint or dizzy spells; severe or untreated exercise-related asthma; or musculoskeletal illness or injury that would be expected to worsen with physical exercise. Additionally, women will be excluded if they are found to have any of the following as measured during the fitness assessment of the first session: a BMI over 40, waist circumference over 40 inches, waist-to-hip ratio of greater than 0.9, systolic blood pressure greater than 150 or diastolic pressure over 95, or resting heart rate over 90.
* factors associated with significant genital nerve damage, including: previous major pelvic surgery that may have caused nerve damage, including hysterectomy, vulvectomy, circumcision, colostomy, cystostomy, or serious bladder, rectal, or abdominal surgery; or neurological impairment due to diabetes, stroke, pelvic nerve damage secondary to trauma, cancer treatments, myasthenia gravis, multiple sclerosis or spinal cord damage.
* factors associated with non-normative endocrine function, including: perimenopausal or menopausal status, or >1 missed menstrual period in the previous 6 months; or currently pregnant, breastfeeding, or having breastfed within the past 3 months; or reporting clinically significant untreated renal or endocrine disease
* untreated serious mental health conditions
* sexual aversion or distress due to history of unwanted sexual contact

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Sexual Functioning | 10 weeks
  Sexual functioning as measured by the Female Sexual Functioning Index

SECONDARY OUTCOMES:
Sexual satisfaction | Baseline (0 weeks), 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks
  Sexual satisfaction as measured by self-report measure completed weekly throughout the trial
Sexual Functioning | 3 weeks, 6 weeks, 9 weeks
  Sexual functioning as measured by the Female Sexual Functioning Index will be measured in between each arm of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Tierney K Lorenz, M.A., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- See also: Laboratory webpage — http://www.mestonlab.com